CLINICAL TRIAL: NCT00741260
Title: A Phase 1/2, Open-Label Study Of Neratinib (HKI-272) In Combination With Capecitabine In Subjects With Solid Tumors And ErbB-2 Positive Metastatic Or Locally Advanced Breast Cancer
Brief Title: Study Evaluating The Combination Of Neratinib And Capecitabine In Solid Tumors And Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-2206 / B1891017
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Solid Tumor; erbB2+ Breast Cancer; Prior trastuzumab; Metastatic; Neratinib; HKI-272; Nerlynx; HER2; PB-272
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — neratinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Neratinib and Capecitabine (Dose Level 1) (Experimental): Neratinib 160 mg and Capecitabine 1500 mg/m^2
  Interventions: Drug: Neratinib; Drug: Capecitabine
- Neratinib and Capecitabine (Dose Group 2) (Experimental): Neratinib 240 mg and Capecitabine 1500 mg/m^2
  Interventions: Drug: Neratinib; Drug: Capecitabine
- Neratinib and Capecitabine (Dose Group 3) (Experimental): Neratinib 240 mg and Capecitabine 2000 mg/m^2
  Interventions: Drug: Neratinib; Drug: Capecitabine
- Neratinib and Capecitabine (Dose Group 4) (Experimental): Neratinib 200 mg and Capecitabine 2000 mg/m^2
  Interventions: Drug: Neratinib; Drug: Capecitabine
- Neratinib and Capecitabine (Dose Group 5) (Experimental): Neratinib 160 mg and Capecitabine 2000 mg/m^2
  Interventions: Drug: Neratinib; Drug: Capecitabine
- Neratinib and Capecitabine MTD (Dose Group 6) (Experimental): Neratinib and Capecitabine Maximum Tolerated Dose without prior lapatinib
  Interventions: Drug: Neratinib; Drug: Capecitabine
- Neratinib and Capecitabine MTD (Dose Group 7) (Experimental): Neratinib and Capecitabine Maximum Tolerated Dose with prior lapatinib
  Interventions: Drug: Neratinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Neratinib — Neratinib orally once daily continually
  Other Names: HKI-272
Drug: Capecitabine — Capecitabine orally on days 1-14 of each 21 day cycle
  Other Names: Xeloda

SUMMARY:
This is a world wide phase 1/2, open-label, study of neratinib in combination with capecitabine, conducted in 2 parts.

In Part 1, 3 to 9 subjects with solid tumors will be enrolled in each dose group of the combination of neratinib and capecitabine. Each subject will participate in only 1 dose group.

Additional subjects may be included at any dose level to further assess the safety and tolerability at that dose level.

In Part 2, up to 60 subjects with erbB-2 positive metastatic breast cancer will receive treatment with the combination of neratinib and capecitabine at the maximum tolerated dose level, as determined in Part 1. In addition 20 subjects with prior lapatinib exposure will be enrolled in Part 2.

Depending on the safety and activity profile observed during the dose escalation phase, the dose selected for Part 2 may be adjusted, if appropriate. In case one test article of the combination is discontinued due to intolerance the other test article can be administered alone.

The primary objectives of Part 1 are to assess the safety and tolerability, and to define the maximum tolerated dose (MTD) of neratinib in combination with capecitabine in subjects with advanced solid tumors.

The primary objective of Part 2 of this study is to confirm the MTD determined in Part 1.

The secondary objective of Part 1 is to collect information on preliminary anti-tumor activity of the combination of neratinib and capecitabine.

Secondary objectives for Part 2 are to collect pharmacokinetic information and to obtain additional efficacy data, such as Objective Response Rate, for subjects with erbB-2 positive breast cancer treated at the MTD of neratinib + capecitabine.

ELIGIBILITY:
INCLUSION CRITERIA

PART 1:

* confirmed pathologic diagnosis of a solid tumor not curable with available therapies for which neratinib plus capecitabine is a reasonable treatment option.

PART 2:

* confirmed histologically and/or cytologically confirmed diagnosis of breast cancer, metastatic or locally advanced.
* erbB-2 gene amplified tumor (FISH or CISH) or erbB-2 overexpression (IHC 3+, or IHC2+ with FISH or CISH confirmation), based on local testing, or based on centralized FISH testing prior to day 1.
* disease progression on or following at least 1 prior trastuzumab containing treatment regimen (at least 6 weeks) for metastatic or locally advanced disease. (Prior adjuvant trastuzumab is allowed but not required). A 2 week period is required between the last dose of trastuzumab treatment and first dose of the test article.
* Prior treatment with a taxane in the neoadjuvant, adjuvant, locally advanced, and/or metastatic disease treatment setting.

PARTS 1 and 2:

* At least 1 measurable lesion as defined by RECIST criteria.
* LVEF within institutional range of normal as measured by multi-gated acquisition (MUGA) or echocardiogram (ECHO).

EXCLUSION CRITERIA

PART 2:

* prior treatment with capecitabine, lapatinib (20 subjects with prior lapatinib exposure will be enrolled) or any erbB-2 targeted agents except trastuzumab. Treatment with erbB-2 targeted therapy must exceed 2 weeks (14 days) in order to be exclusionary.
* prior treatment with anthracyclines with a cumulative dose of doxorubicin of greater than 400 mg/m², epirubicin dose of greater than 800 mg/m², or the equivalent dose for other anthracyclines.

PARTS 1 and 2:

* Subjects with bone as the only site of disease.
* Active uncontrolled or symptomatic central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Subjects with a history of CNS metastases or cord compression are allowable if they have been considered definitively treated and are off anticonvulsants and steroids for at least 4 weeks before the first dose of test article.
* Any other cancer within 5 years prior to screening with the exception of adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-12-09 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (37):
- United States (12):
  - USA Mitchell Cancer Institute, Mobile, Alabama
  - Pacific Shores Medical Group, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Kootenai Cancer Center, Post Falls, Idaho
  - The Care Group, LLC. dba Horizon Oncology Center, Lafayette, Indiana
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Arena Oncology Associates, PC, Lake Success, New York
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Berks Hematology Oncology, West Reading, Pennsylvania
  - HOPE Oncology, Richardson, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center Institute for Drug Development, San Antonio, Texas
- Australia (2):
  - Mater Private Centre for HOCA, South Brisbane, Queensland
  - Border Medical Oncology, Wodonga, Victoria
- Brazil (2):
  - Associacao Hospitalar Moinhos de Vento Instituto de Edicacao e Pesquisa, Porto Alegre, Rio Grande do Sul
  - Associacao Hospital de Caridade Ijui, Ijuí, RS - Brazil
- China (4):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The Hospital Affiliated Academy Military Medical Science, Chinese People's Liberation Army, Beijing
- University Hospital Center Zagreb Department of Oncology, Zagreb, Croatia
- UNIMED Medical Institute, Comprehensive Centre for Breast Diseases, Hong Kong, Hong Kong
- Hungary (2):
  - Orszagos Onkologiai Intezet "B" Belgyogyaszati osztaly, Budapest
  - Josa Andras Oktatokorhaz / Onkoradiologiai Osztaly, Nyíregyháza
- Russia (5):
  - Republican Clinical Oncology Dispensary, Kazan'
  - GUZ Perm Regional Oncology Dispensary, Perm
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - GUZ City Clinical Oncology Dispensary, Saint Petersburg
  - Saint-Petersburg State Medical University n.a. acad. I.P. Pavlov, Laboratory of Thoracic Oncology of Pulmonology Research Institute, Saint Petersburg
- Johns Hopkins Singapore International Medical Centre, Singapore, Singapore
- South Korea (3):
  - Yonsei University Health System-Severance Hospital, Yonsei University College of Medicine, Seoul
  - Department of Hematology/Oncology, Samsung Medical Center, Seoul
  - Asan Medical Center Department of Medicine Division of Oncology, Seoul
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Saura C, Garcia-Saenz JA, Xu B, Harb W, Moroose R, Pluard T, Cortes J, Kiger C, Germa C, Wang K, Martin M, Baselga J, Kim SB. Safety and efficacy of neratinib in combination with capecitabine in patients with metastatic human epidermal growth factor receptor 2-positive breast cancer. J Clin Oncol. 2014 Nov 10;32(32):3626-33. doi: 10.1200/JCO.2014.56.3809. Epub 2014 Oct 6. PMID 25287822

RESULTS

PARTICIPANT FLOW:
Groups:
- N160 + C1500: Neratinib 160 mg + Capecitabine 1500 mg/sq m
- N240 + C1500: Neratinib 240 mg + Capecitabine 1500 mg/sq m
- N240 + C2000: Neratinib 240 mg + Capecitabine 2000 mg/sq m
- N200 + C2000: Neratinib 200 mg + Capecitabine 2000 mg/sq m
- N160 + C2000: Neratinib 160 mg + Capecitabine 2000 mg/sq m
- N + C MTD - No Prior Lap: Neratinib + Capecitabine MTD (No prior Lapatinib)
- N + C MTD - Prior Lap: Neratinib + Capecitabine MTD (Prior Lapatinib)
Period: Overall Study
Arm/Group | N160 + C1500 | N240 + C1500 | N240 + C2000 | N200 + C2000 | N160 + C2000 | N + C MTD - No Prior Lap | N + C MTD - Prior Lap
Started | 6 | 8 | 4 | 6 | 9 | 65 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 20 | 0
Not Completed | 6 | 8 | 4 | 6 | 9 | 45 | 7
Not completed — Disease Progression | 3 | 5 | 3 | 3 | 5 | 37 | 4
Not completed — Death | 0 | 1 | 0 | 1 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 3 | 1
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 1 | 2 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | N160 + C1500 | N240 + C1500 | N240 + C2000 | N200 + C2000 | N160 + C2000 | N + C MTD - No Prior Lap | N + C MTD - Prior Lap | Total
Number analyzed (Participants) | 6 | 8 | 4 | 6 | 9 | 65 | 7 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 3 | 3 | 7 | 59 | 7 | 91
  >=65 years | 1 | 1 | 1 | 3 | 2 | 6 | 0 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.50) | 53.3 (10.42) | 56.3 (17.15) | 59.0 (10.88) | 55.7 (10.64) | 51.5 (10.48) | 50.9 (10.65) | 52.4 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 3 | 6 | 65 | 7 | 93
  Male | 2 | 3 | 1 | 3 | 3 | 0 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 25 | 3 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
  White | 5 | 8 | 4 | 6 | 9 | 38 | 4 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Number of participants reporting Adverse Events Causing Dose Limiting Toxicities (DLT).
Time Frame: From first dose date to day 21
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- N160 + C1500: Neratinib 160 mg + Capecitabine 1500 mg/m2
- N160 + C2000: Neratinib 160 mg + Capecitabine 2000 mg/m2
- N200 + C2000: Neratinib 200 mg + Capecitabine 2000 mg/m2
- N240 + C1500: Neratinib 240 mg + Capecitabine 1500 mg/m2
- N240 + C2000: Neratinib 240 mg + Capecitabine 2000 mg/m2
Arm/Group | N160 + C1500 | N160 + C2000 | N200 + C2000 | N240 + C1500 | N240 + C2000 | N + C MTD - No Prior Lap | N + C MTD - Prior Lap
Number analyzed (Participants) | 6 | 9 | 6 | 8 | 4 | 65 | 7
Participants | 0 | 2 | 2 | 0 | 2 | 0 | 0

2. Secondary Outcome: Overall Response Rate
Description: Number of Subjects with Complete or Partial Response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression or last tumor assessment, up to three years.
Population: Evaluable Population includes subjects who met all inclusion/exclusion criteria, received at least two weeks of neratinib and capecitabine, and underwent valid tumor assessments at baseline and at least one post-baseline time point stratified by prior Lapatinib exposure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Prior Lapatinib Subjects: MTD (Part 2), Subjects with Prior Lapatinib Experience
- Lapatinib Naive Subjects P1: MTD (Part 2), Subjects without Prior Lapatinib Experience
- Lapatinib Naive Subjects Part 2 + Part 1: MTD (Part 2 + Part 1), Subjects without Prior Lapatinib Experience
Arm/Group | Prior Lapatinib Subjects | Lapatinib Naive Subjects P1 | Lapatinib Naive Subjects Part 2 + Part 1
Number analyzed (Participants) | 7 | 61 | 63
percentage of participants | 57.1 [18.4 to 90.1] | 63.9 [50.6 to 75.8] | 63.5 [50.4 to 75.3]

3. Secondary Outcome: Clinical Benefit Rate
Description: The percentage of subjects with Complete Response, Partial Response, or Stable Disease at least 24 weeks per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From first dose date to progression or last tumor assessment, up to three years.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior Lapatinib Subjects | Lapatinib Naive Subjects P1 | Lapatinib Naive Subjects Part 2 + Part 1
Number analyzed (Participants) | 7 | 61 | 63
percentage of participants | 71.4 [29.0 to 96.3] | 72.1 [59.2 to 82.9] | 73.0 [60.3 to 83.4]

4. Secondary Outcome: Duration of Response
Description: Duration of response was measured from the time at which response criteria were met for complete response (CR) or partial response (PR) (whichever status was recorded first) until the first date of recurrence or progressive disease (PD) or death per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From start date of response to first PD/death, up to three years.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Prior Lapatinib Subjects | Lapatinib Naive Subjects P1 | Lapatinib Naive Subjects Part 2 + Part 1
Number analyzed (Participants) | 4 | 39 | 40
weeks | 48.3 [30.0 to 61.0] | 46.3 [30.1 to NA] — Upper limit of the 95% confidence interval not estimable due to insufficient number of participants with events. | 46.3 [30.1 to NA] — Upper limit of the 95% confidence interval not estimable due to insufficient number of participants with events.

5. Primary Outcome: Maximum Tolerated Dose (MTD) of Neratinib
Description: MTD reflects the highest dose of neratinib plus capeciteabine that did not cause a selected Grade 3 toxicity in >= 2 participants, which is any of 1) Grade 3 or 4 non-hematologic toxicity (Grade 3 asthenia was not considered a DLT unless lasting >3 days, 2) Grade 3 diarrhea lasting >2 days on optimal medical therapy or associated with fever or dehydration. 3) Grade 4 neutropenia lasting ≥ 3 days or Grade 4 febrile neutropenia, 4) Grade 4 thrombocytopenia lasting ≥3 days or associated with bleeding or requiring platelet transfusion, 5) Delayed recovery [to ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or baseline] from one of the above listed toxicities that were related to neratinib and/or capecitabine that delayed the initiation of the next dose by more than 3 weeks.
Time Frame: From first dose date to day 21.
Population: All patients in the safety population in part 1 (dose-escalation) of the study.
Measure: Number; unit: mg
Groups:
- Neratinib in Combination With Capecitabine: Oral Neratinib administered daily in combination with capecitabine orally on days 1-14 of each 21 day cycle
Arm/Group | Neratinib in Combination With Capecitabine
Number analyzed (Participants) | 33
mg | 240

6. Primary Outcome: Maximum Tolerated Dose (MTD) of Capecitabine
Description: MTD reflects the highest dose of capecitabine in combination with neratinib that did not cause a selected Grade 3 toxicity in >= 2 participants, which is any of 1) Grade 3 or 4 non-hematologic toxicity (Grade 3 asthenia was not considered a DLT unless lasting >3 days, 2) Grade 3 diarrhea lasting >2 days on optimal medical therapy or associated with fever or dehydration. 3) Grade 4 neutropenia lasting ≥ 3 days or Grade 4 febrile neutropenia, 4) Grade 4 thrombocytopenia lasting ≥3 days or associated with bleeding or requiring platelet transfusion, 5) Delayed recovery [to ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or baseline] from one of the above listed toxicities that were related to neratinib and/or capecitabine that delayed the initiation of the next dose by more than 3 weeks.
Time Frame: From first dose date to day 21.
Population: All patients in the safety population in part 1 (dose-escalation) of the study.
Measure: Number; unit: mg/m^2
Groups:
- Capecitabine in Combination With Neratinib: Oral Neratinib administered daily in combination with capecitabine orally on days 1-14 of each 21 day cycle
Arm/Group | Capecitabine in Combination With Neratinib
Number analyzed (Participants) | 33
mg/m^2 | 1500

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, up to five years.
Arm/Group | N160 + C1500 | N240 + C1500 | N240 + C2000 | N200 + C2000 | N160 + C2000 | N + C MTD - No Prior Lap | N + C MTD - Prior Lap
Serious Adverse Events (participants affected / at risk) | 5/6 | 4/8 | 2/4 | 3/6 | 3/9 | 19/65 | 2/7
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 4/4 | 6/6 | 9/9 | 62/65 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N160 + C1500 (N=6) | N240 + C1500 (N=8) | N240 + C2000 (N=4) | N200 + C2000 (N=6) | N160 + C2000 (N=9) | N + C MTD - No Prior Lap (N=65) | N + C MTD - Prior Lap (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Biloma (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N160 + C1500 (N=6) | N240 + C1500 (N=8) | N240 + C2000 (N=4) | N200 + C2000 (N=6) | N160 + C2000 (N=9) | N + C MTD - No Prior Lap (N=65) | N + C MTD - Prior Lap (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 11 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 8 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 5 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 8 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 7 | 4 | 6 | 8 | 59 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 11 | 2
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 3 | 3 | 25 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 12 | 0
Vomiting (Gastrointestinal disorders) | 1 | 6 | 2 | 1 | 3 | 21 | 3
Asthenia (General disorders) | 2 | 4 | 2 | 2 | 5 | 12 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 1 | 1 | 4 | 15 | 2
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Implant site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Injection site extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 3 | 1 | 2 | 0 | 9 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0
Pyrexia (General disorders) | 2 | 2 | 1 | 1 | 2 | 6 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 8 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 9 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 4 | 0
Wound infection pseudomonas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 1 | 2 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 1 | 2 | 11 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 1 | 2 | 10 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 3 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 6 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 6 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0 | 2 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 7 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 4 | 2 | 19 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1 | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1 | 0 | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 8 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 7 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 12 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0 | 3 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 0 | 0 | 0 | 9 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 10 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 5 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 7 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 1 | 4 | 41 | 5
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 13 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less